CLINICAL TRIAL: NCT01276704
Title: Flaxseed Lignan as a Prevention Strategy for Pre-Menopausal Women at High Risk for Development of Breast Cancer
Brief Title: Prevention Strategy for Pre-Menopausal Women at High Risk for Development of Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual rate lower than anticipated; funding expired
Sponsor: Carol Fabian, MD (Other)
Collaborators: Lignan Research Inc. (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12377
Record Dates: First submitted 2011-01-06; First posted 2011-01-13 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — secoisolariciresinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flaxseed lignan, SDG (Experimental): Secoisolariciresinol diglycoside
  Interventions: Drug: secoisolariciresinol
- Placebo (Placebo Comparator): Matched Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — The placebo contains same filler materials as commercially available Brevail® but without active SDG.
  Arms: Placebo
Drug: secoisolariciresinol — 1 capsule daily of secoisolariciresinol diglycoside (SDG)50mg
  Other Names: SDG
  Arms: flaxseed lignan, SDG

SUMMARY:
The investigators will study the effect of 12 months of SDG (Brevail) vs placebo on women at increased risk for development of breast cancer.

DETAILED DESCRIPTION:
The investigators would like to see if women at increased risk for breast cancer are likely to tolerate SDG daily for 12 months without significant side effects or changes in their menstrual cycles. The investigators would also like to determine if Brevail® can reduce breast cell proliferation in pre-menopausal women.

ELIGIBILITY:
PARTICIPANT SELECTION

* Risk Level Required for RPFNA Screening for Eligibility

  * Given the low probability of side effects and the desire to be able to generalize results to a moderate as well as high risk population, the target cohort is pre-menopausal women who have a relative risk for breast cancer which is 2-fold or greater than that of the average woman in their age group by virtue of any one of the following conditions:
* A 1st or 2nd degree relative with breast cancer diagnosed under the age of 60
* A prior biopsy indicating proliferative breast disease, atypical hyperplasia, or LCIS
* Multiple prior breast biopsies regardless of histology
* 50% or higher estimated mammographic density on visual inspection
* Prior or current RPFNA evidence of atypia
* Known carrier of a BRCA1 or 2 mutation.

  * Age, Life-Style and Medical Eligibility Criteria for Tissue Screening

Candidates for tissue screening for this study are pre-menopausal women who meet the risk criteria above and all of the following demographic and medical criteria:

* Age 21 to 49 (limiting the maximum age to 49 will reduce the possibility of reduction in Ki-67 due to entry into menopause transition during the study).
* Stable hormonal status for the previous 6 months (has not stopped or started oral contraceptives, or experienced lactation or pregnancy) and willing to maintain same status while on study.
* BMI < 40 kg/m2.
* Has had at least 4 menstrual cycles in past year
* If regularly undergoing screening mammography, must have been performed within 9 months prior to baseline RPFNA, and interpreted as not suspicious for breast cancer
* Breast exam interpreted as normal (not suspicious for cancer).

  * Exclusion Criteria for Screening RPFNA and Study Participation

Candidates are ineligible for tissue screening if they meet any of the following conditions:

* Consumption of systemic antibiotics during the 3 weeks prior to baseline RPFNA. Systemic antibiotics reduce intestinal bacteria and thus the ability to convert SECO to ENL.
* Consumption of supplements containing SDG (flaxseed or sesame seed) during the 3 weeks prior to baseline RPFNA. ( Consumption of foods containing flaxseed or sesame seed are OK.)
* Use of any selective estrogen receptor modulator or aromatase inhibitor (tamoxifen, raloxifene, arzoxifene, acolbifene, anastrozole, exemestane, letrozole) within the previous 6 months.
* Currently enrolled on an interventional investigational study.
* Bilateral breast implants.
* Invasive breast cancer or other invasive cancer diagnosis within five years.
* Metastatic malignancy of any kind.excluding Hodgkin's or non-Hodgkin's lymphoma.
* Current anticoagulant use.
* Consumption of coumadin, fish oil, or other anticoagulants during the 3 weeks prior to baseline RPFNA.
* Any other condition or intercurrent illness that in the opinion of the investigator makes the subject a poor candidate for RPFNA or the trial.

  * Inclusion Criteria for Study Entry
* RPFNA performed in the follicular portion (day 1-10) of the menstrual cycle. Note that day 1 is defined as the first day of bleeding.
* RPFNA specimen exhibits hyperplasia +/- atypia (Masood score of ≥13) with ≥500 cells on the cytology slide.
* Ki-67 ≥2% positivity (≥500 cells).
* Willing to continue without oral contraceptives throughout the duration of the study participation (12 months). Non-oral contraceptives are permissible. If heterosexually active, must be agreeable to use some non-hormonal form of contraception during the trial or husband or partner must have had a vasectomy. (Safety of SDG during pregnancy has not been documented).
* Have reasonable organ function as documented by metabolic chemistry profile.
* Willing to undergo a history and physical at baseline and 12 months and be contacted periodically by the trial coordinator during the 12 month study period.
* Willing to have blood drawn at baseline and twelve months.
* Able to understand and willing to provide informed consent for the RPFNA's and study participation.

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (7):
- United States (7):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Ohio State Unviersity Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Global results will be published.

REFERENCES:
- [Result] Fabian CJ, Khan SA, Garber JE, Dooley WC, Yee LD, Klemp JR, Nydegger JL, Powers KR, Kreutzjans AL, Zalles CM, Metheny T, Phillips TA, Hu J, Koestler DC, Chalise P, Yellapu NK, Jernigan C, Petroff BK, Hursting SD, Kimler BF. Randomized Phase IIB Trial of the Lignan Secoisolariciresinol Diglucoside in Premenopausal Women at Increased Risk for Development of Breast Cancer. Cancer Prev Res (Phila). 2020 Jul;13(7):623-634. doi: 10.1158/1940-6207.CAPR-20-0050. Epub 2020 Apr 20. PMID 32312713

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 180 participants were screened and found to be eligible. Two withdrew consent prior to being randomized. Of the 178 randomized, 116 were assigned to active agent; 62 to placebo. One active agent participant withdrew prior to receiving study agent. The 177 who received study agent constitute the analytic population.
Period: Overall Study
Arm/Group | Flaxseed Lignan, SDG | Placebo
Started | 115 | 62
Completed | 101 | 51
Not Completed | 14 | 11
Not completed — Lost to Follow-up | 2 | 3
Not completed — Non-compliant | 2 | 2
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Physician Decision | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flaxseed Lignan, SDG | Placebo | Total
Number analyzed (Participants) | 115 | 62 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (6.7) | 39.7 (6.1) | 38.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 62 | 177
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 108 | 60 | 168
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 103 | 59 | 162
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 115 | 62 | 177
Ki-67 expression [Mean (Standard Deviation); unit: percent of breast epithelial cells] — Percent of breast epithelial cells expressing Ki-67 assessed immunocytochemically.
  percent of breast epithelial cells | 6.1 (0.4) | 5.4 (4.2) | 5.9 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Breast Epithelial Cells With Ki-67 Immunocytochemical Expression
Description: Change over the course of study in the percent of breast epithelial cells expressing the proliferation marker Ki- 67/MIB-1 in hyperplastic benign breast tissue acquired by random periareolar fine needle aspiration pre-study and post-study.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: change in percent Ki-67
Arm/Group | Flaxseed Lignan, SDG | Placebo
Number analyzed (Participants) | 101 | 51
change in percent Ki-67 | -1.4 (5.3) | -1.4 (5.3)
Statistical Analysis 1: Comparison: Flaxseed Lignan, SDG vs Placebo; 83% power to detect an absolute 2.5% reduction in Ki-67 for the treatment group compared with no reduction in the control group; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance: < 0.05

2. Secondary Outcome: Change in Gene Expression
Description: Gene expression in breast epithelial cells assessed by RT-qPCR. Change in expression (fold-change for 12-months compared to baseline value) was evaluated by cluster analysis and used to define "responders" and non-responders" based on favorable or non-favorable modulation of a set of 12 relevant genes.
  Specifically, data for change in ESR1 (codes for estrogen receptor alpha) are shown.
Time Frame: 12 months
Population: Adequate residual material available from baseline and 12-month specimens for post-hoc analysis of change in gene expression.
Measure: Count of Participants; unit: Participants
Arm/Group | Flaxseed Lignan, SDG | Placebo
Number analyzed (Participants) | 49 | 28
Participants
  > 2-fold increase | 3 | 7
  No substantial change | 36 | 19
  < 0.5 fold change | 10 | 2
Statistical Analysis 1: Comparison: Flaxseed Lignan, SDG vs Placebo; Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. Standard threshold of P<0.05

3. Secondary Outcome: Breast Cancer Prevention Trial (BCPT) Symptom Checklist
Description: Quality of life as measured by the Breast Cancer Prevention Trial (BCPT) Symptom Checklist, completed at baseline and end of study by each participant.
  Responses to 43 questions (with each question given a value from 0 to 4, higher score being worse) are clustered into seven domains to yield an average score per domain. These seven category scores are then averaged to provide a final average score (range by definition, 0 to 4). Change in score over the course of the intervention per individual is then assessed. By definition, change in score theoretically ranges from -4 to +4.
Time Frame: 12 months
Measure: Median (Full Range); unit: Change in score on a scale
Arm/Group | Flaxseed Lignan, SDG | Placebo
Number analyzed (Participants) | 101 | 51
Change in score on a scale | -0.05 [-2.3 to 1.4] | 0.21 [-1.4 to 2.7]
Statistical Analysis 1: Comparison: Flaxseed Lignan, SDG vs Placebo; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. Standard threshold of P < 0.05

ADVERSE EVENTS:
Time Frame: 12 months
Description: When individual (non-serious) adverse events are diverse, with small numbers in any one event type, total numbers of participants reporting the most severe AE grade are reported.
Arm/Group | Flaxseed Lignan, SDG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/115 | 4/62
Other Adverse Events (participants affected / at risk) | 84/115 | 45/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flaxseed Lignan, SDG (N=115) | Placebo (N=62)
vestibular disorder (Nervous system disorders) | 0 (0) | 1 (1) — diagnosis of vestibular schwannoma (grade 2)
musculoskeletal connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — diagnosis of desmoid tumor (grade 3)
sinus disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) — septoplasty for a deviated septum (grade 3)
Breast abnormality (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — diagnosis of DCIS (grade 3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 3
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — miscarriage requiring a D&C procedure (grade 5 for fetal death).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flaxseed Lignan, SDG (N=115) | Placebo (N=62)
Grade 1 AE (Product Issues) | 36 (36) | 17 (17) — Total number of participants reporting a grade 1 AE.
Grade 2 AE (Product Issues) | 39 (39) | 24 (24) — Total number of participants reporting a grade 2 AE.
Grade 3 AE (Product Issues) | 9 (9) | 8 (8) — Total number of participants reporting a grade 3 AE.

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed. A total of 240 enrollees was planned; actual accrual was 180.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT01276704/Prot_SAP_000.pdf